CLINICAL TRIAL: NCT03929393
Title: Mindful Movement for Physical Activity and Wellbeing in Older Adults- A Community Based Randomized Hybrid Effectiveness-Implementation Study
Brief Title: Mindful Movement for Physical Activity and Wellbeing in Older Adults- A Hybrid Effectiveness-Implementation Study
Acronym: Y-U
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: YMCA (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1611S99323; R33AT009110 (NIH)
Record Dates: First submitted 2019-04-16; First posted 2019-04-26 (Actual); Results first posted 2023-07-21 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Physical Inactivty; Wellbeing; Mindfulness
Keywords: Randomized controlled trial; Exercise; Physical Activity; Behavior Change; Mindfulness; Aging
MeSH Terms: conditions — Motor Activity | interventions — Health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Movement (Experimental): 8, 90-minute, in-person, group sessions over 8 weeks
  Interventions: Behavioral: Mindful Movement
- Keys to Health & Wellbeing (Active Comparator): 8, 90-minute, in-person, group sessions over 8 weeks
  Interventions: Other: Keys to Health & Wellbeing

INTERVENTIONS:
Behavioral: Mindful Movement — The program focuses on enhancing individuals' mindfulness capabilities and skills, specifically attention regulation, body awareness, emotional regulation, and shifts in self-perception, by providing opportunities for education, practice, and social suppo
  Arms: Mindful Movement
Other: Keys to Health & Wellbeing — This community-based educational program provides participants useful content focused on general health related topics including common chronic conditions, social support, social participation, cancer screening, immunization and keeping active.
  Arms: Keys to Health & Wellbeing

SUMMARY:
Physical inactivity has reached pandemic proportions and is associated with increased morbidity, mortality, and healthcare costs. Of particular concern is that most middle to older age adults fall far short of recommendations for health enhancing physical activities. This research takes a novel approach to tackling this problem by combining mindfulness with behavioral strategies in a unique 'Mindful Movement' program offered collaboratively with the YMCA.

ELIGIBILITY:
Inclusion Criteria:

≥ 50 years of age

* Accelerometer wear time ≥10 hours on at least 4 days in a 7 consecutive day period between baselines
* Self-report of <140 minutes of MVPA per week in 3 months prior to baseline AND accelerometer recorded <100 minutes of MVPA between baselines
* Mini-Mental State score ≥ 24 if indicated
* Independent self-ambulation
* Provides consent and is willing to participate in data collection activities

Exclusion Criteria:

* Pregnancy
* Unwilling or unable to participate in study activities
* Current or upcoming participation in educational programs similar to those under study
* Medical restrictions to increasing Moderate Vigorous Physical Activity (MVPA)
* Terminal illness
* Contraindications to mindfulness practice

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - YMCA Burnsville, Burnsville, Minnesota
  - YMCA Southdale, Edina, Minnesota
  - YMCA Cora McCorvey, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - YMCA Midway, Saint Paul, Minnesota

REFERENCES:
- See also: Study Website — https://csh.umn.edu/research/nih-y-u-research-study

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindful Movement: 8, 90-minute, in-person, group sessions over 8 weeks
  The program focuses on enhancing individuals' mindfulness capabilities and skills, specifically attention regulation, body awareness, emotional regulation, and shifts in self-perception by providing opportunities for education, practice, and social support.
Period: Overall Study
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Started | 86 | 90
Completed | 82 | 80
Not Completed | 4 | 10
Not completed — Death | 1 | 0
Not completed — Time Commitment | 2 | 5
Not completed — Motor Vehicle Accident | 0 | 1
Not completed — Difficulty Using Videoconferencing Technology | 0 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindful Movement | Keys to Health & Wellbeing | Total
Number analyzed (Participants) | 86 | 90 | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (7.2) | 66.8 (8.4) | 66.2 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 74 | 152
  Male | 8 | 16 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 82 | 85 | 167
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 8 | 12
  White | 75 | 80 | 155
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 86 | 90 | 176

OUTCOME MEASURES:

1. Primary Outcome: Moderate-Vigorous Physical Activity (MVPA) in 10 Min Bouts
Description: Minutes/week spent in ≥10-min bouts of MVPA
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 18.35 (24.97) | 15.54 (23.94)

2. Primary Outcome: Moderate-Vigorous Physical Activity (MVPA) in 10 Min Bouts
Description: Minutes/week spent in ≥10-min bouts of MVPA
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 39.5 [24.5 to 57.5] | 24.3 [12.6 to 35.7]

3. Secondary Outcome: Moderate-Vigorous Physical Activity (MVPA) in 10 Min Bouts
Description: Minutes/week spent in ≥10-min bouts of MVPA
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 28.0 [14.5 to 44.0] | 16.2 [8.4 to 24.9]

4. Secondary Outcome: Moderate-Vigorous Physical Activity (MVPA) in 10 Min Bouts
Description: Minutes/week spent in ≥10-min bouts of MVPA
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 20.7 [10.7 to 32.5] | 11.3 [3.4 to 20.4]

5. Secondary Outcome: Total Moderate-Vigorous Physical Activity (MVPA)
Description: Minutes/week spent in MVPA
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 91.9 (74.3) | 93.0 (95.2)

6. Secondary Outcome: Total Moderate-Vigorous Physical Activity (MVPA)
Description: Minutes/week spent in MVPA
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 49.2 [29.0 to 69.4] | 34.4 [14.5 to 54.3]

7. Secondary Outcome: Total Moderate-Vigorous Physical Activity (MVPA)
Description: Minutes/week spent in MVPA
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 43.0 [23.4 to 62.7] | 23.1 [3.8 to 42.5]

8. Secondary Outcome: Total Moderate-Vigorous Physical Activity (MVPA)
Description: Minutes/week spent in MVPA
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 20.6 [1.0 to 40.2] | 8.8 [-10.5 to 28.0]

9. Secondary Outcome: Sedentary Activity
Description: Time spent in sedentary activity
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 2804 (912) | 2988 (1069)

10. Secondary Outcome: Sedentary Activity
Description: Time spent in sedentary activity
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | -85 [-256 to 85] | -46 [-214 to 123]

11. Secondary Outcome: Sedentary Activity
Description: Time spent in sedentary activity
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | -246 [-432 to -60] | -209 [-392 to -26]

12. Secondary Outcome: Sedentary Activity
Description: Time spent in sedentary activity
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 51 [-137 to 238] | 153 [-31 to 336]

13. Secondary Outcome: Average Daily Step Count
Description: Average steps/day over one week
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: steps per day
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
steps per day | 3694 (1753) | 3217 (1595)

14. Secondary Outcome: Average Daily Step Count
Description: Average steps/day over one week
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
steps per day | 831 [479 to 1182] | 754 [408 to 1100]

15. Secondary Outcome: Average Daily Step Count
Description: Average steps/day over one week
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
steps per day | 1100 [733 to 1467] | 849 [488 to 1210]

16. Secondary Outcome: Average Daily Step Count
Description: Average steps/day over one week
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
steps per day | 476 [111 to 842] | 96 [-263 to 455]

17. Secondary Outcome: Quality of Life - Euroqol 5D (EQ5D)
Description: The EQ5D captures five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) over 5 levels (no problem, slight problem, moderate problem, severe problem, unable to perform/extreme problem). The scale for the EQ5D ranges from -0.109 to 1, with higher scores indicating higher quality of life.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.89 (0.12) | 0.89 (0.12)

18. Secondary Outcome: Quality of Life - Euroqol 5D (EQ5D)
Description: as for outcome 17
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -0.03 [-0.06 to -0.03] | -0.05 [-0.08 to -0.03]

19. Secondary Outcome: Quality of Life - Euroqol 5D (EQ5D)
Description: as for outcome 17
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -0.06 [-0.08 to -0.03] | -0.06 [-0.09 to -0.04]

20. Secondary Outcome: Quality of Life - Euroqol 5D (EQ5D)
Description: as for outcome 17
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -0.05 [-0.08 to -0.03] | -0.07 [-0.10 to -0.04]

21. Secondary Outcome: Quality of Life - EuroQol VAS
Description: The EuroQol VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement. Results are on a 0 to 100 scale with higher scores indicating better self-rated health.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 75.3 (14.6) | 74.0 (13.3)

22. Secondary Outcome: Quality of Life - EuroQol VAS
Description: as for outcome 21
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 2.1 [-0.6 to 4.8] | -1.0 [-3.6 to 1.7]

23. Secondary Outcome: Quality of Life - EuroQol VAS
Description: as for outcome 21
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -0.7 [-3.6 to 2.1] | -0.9 [-3.6 to 1.9]

24. Secondary Outcome: Quality of Life - EuroQol VAS
Description: as for outcome 21
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.0 [-2.9 to 2.9] | 1.1 [-1.7 to 3.9]

25. Secondary Outcome: Exercise Self-Efficacy- Self-Efficacy for Exercise (SEE) Scale
Description: Individuals are asked to rate their confidence in their ability to exercise. Confidence ratings range from 0 (not confident) to 10 (very confident). The average of all responses is used for a total score ranging from 0 to 10. Higher scores indicate higher exercise self-efficacy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 7.8 (1.8) | 7.0 (2.5)

26. Secondary Outcome: Exercise Self-Efficacy- Self-Efficacy for Exercise (SEE) Scale
Description: as for outcome 25
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -1.8 [-2.3 to -1.3] | -1.6 [-2.1 to -1.1]

27. Secondary Outcome: Exercise Self-Efficacy- Self-Efficacy for Exercise (SEE) Scale
Description: as for outcome 25
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -1.8 [-2.3 to -1.3] | -1.6 [-2.1 to -1.1]

28. Secondary Outcome: Exercise Self-Efficacy- Self-Efficacy for Exercise (SEE) Scale
Description: as for outcome 25
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | -2.0 [-2.6 to -1.4] | -1.8 [-2.4 to -1.2]

29. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Positive Sub-scale
Description: This is a 13-item instrument focused on beliefs about the positive and negative physical and mental health benefits of exercise. The OEE-2 includes positive and negative outcome expectations sub-scales. Responses range from 1 (strongly agree) to 5 (strongly disagree) and are averaged with final scores ranging from 1 to 5. Lower scores indicate stronger exercise expectations.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.6 (0.5) | 1.7 (0.5)

30. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Positive Sub-scale
Description: as for outcome 29
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.0 [-0.1 to 0.1] | 0.1 [0.0 to 0.2]

31. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Positive Sub-scale
Description: as for outcome 29
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.0 [-0.1 to 0.1] | 0.1 [0.0 to 0.2]

32. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Positive Sub-scale
Description: as for outcome 29
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.1 [0.0 to 0.2] | 0.1 [0.0 to 0.3]

33. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Negative Sub-scale
Description: as for outcome 29
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.5 (0.6) | 1.8 (0.6)

34. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Negative Sub-scale
Description: as for outcome 29
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.2 [0.0 to 0.3] | 0.1 [-0.1 to 0.2]

35. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Negative Sub-scale
Description: as for outcome 29
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.1 [0.0 to 0.3] | 0.2 [0.0 to 0.3]

36. Secondary Outcome: Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) Negative Sub-scale
Description: as for outcome 29
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.2 [0.0 to 0.3] | 0.2 [0.1 to 0.4]

37. Secondary Outcome: Mindfulness - Mindful Attention Awareness Scale (MAAS)
Description: The MAAS scale is comprised of 15 items measured on a 6-point scale (1=almost always, 6=almost never). Responses to individual items are averaged for a total scale ranging from 1 to 6. Higher scores indicate stronger dispositional mindfulness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 4.2 (0.9) | 4.4 (0.8)

38. Secondary Outcome: Mindfulness - Mindful Attention Awareness Scale (MAAS)
Description: as for outcome 37
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.0 [-0.1 to 0.1] | 0.0 [-0.2 to 0.1]

39. Secondary Outcome: Mindfulness - Mindful Attention Awareness Scale (MAAS)
Description: as for outcome 37
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.2 [0.0 to 0.3] | 0.1 [0.0 to 0.2]

40. Secondary Outcome: Mindfulness - Mindful Attention Awareness Scale (MAAS)
Description: as for outcome 37
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.2 [0.0 to 0.3] | 0.0 [-0.1 to 0.2]

41. Secondary Outcome: Mindfulness - Frieberg Mindfulness Inventory (FMI)
Description: The FMI addresses 14 items with a four-point response scale (1=rarely, 4=almost always). Items are summed scores ranging from 14 to 56. Higher scores indicate more mindfulness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 37.3 (7.9) | 38.5 (7.0)

42. Secondary Outcome: Mindfulness - Frieberg Mindfulness Inventory (FMI)
Description: as for outcome 41
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 3.4 [2.2 to 4.6] | 0.3 [-0.9 to 1.4]

43. Secondary Outcome: Mindfulness - Frieberg Mindfulness Inventory (FMI)
Description: as for outcome 41
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 3.2 [1.8 to 4.6] | 1.1 [-0.3 to 2.4]

44. Secondary Outcome: Mindfulness - Frieberg Mindfulness Inventory (FMI)
Description: as for outcome 41
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 3.5 [2.1 to 5.0] | 0.7 [-0.7 to 2.1]

45. Secondary Outcome: Wellbeing-8-item Flourishing Scale
Description: This 8 item scale assesses perceived success in relationships, self-esteem, and purpose. Responses are 7=Strongly Agree to 1=Strongly Disagree. The total score ranges from 8 to 56. Higher scores indicate better perceived wellbeing.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 45.7 (7.0) | 46.0 (6.0)

46. Secondary Outcome: Wellbeing-8-item Flourishing Scale
Description: as for outcome 45
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.3 [0.2 to 2.4] | 0.3 [-0.7 to 1.4]

47. Secondary Outcome: Wellbeing-8-item Flourishing Scale
Description: as for outcome 45
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.8 [-0.4 to 2.0] | 0.6 [-0.6 to 1.8]

48. Secondary Outcome: Wellbeing-8-item Flourishing Scale
Description: as for outcome 45
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.3 [0.0 to 2.5] | 0.1 [-1.1 to 1.4]

49. Secondary Outcome: Social Connectedness
Description: Eight-item questionnaire with responses ranging from 1=strongly agree to 6=strongly disagree. Items are summed with the total scale ranging from 8 to 48. Higher scores indicates more social connectedness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 40.1 (7.5) | 41.7 (6.5)

50. Secondary Outcome: Social Connectedness
Description: as for outcome 49
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.4 [0.1 to 2.7] | -0.6 [-1.9 to 0.7]

51. Secondary Outcome: Social Connectedness
Description: as for outcome 49
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.0 [-0.5 to 2.4] | -1.1 [-2.5 to 0.3]

52. Secondary Outcome: Social Connectedness
Description: as for outcome 49
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.2 [-0.3 to 2.7] | -0.9 [-2.3 to 0.5]

53. Secondary Outcome: Social Assuredness
Description: Eight-item questionnaire with responses ranging from 1=strongly agree to 6=strongly disagree. Items are summed with the total scale ranging from 8 to 48. Higher scores indicates more social assuredness or confidence.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 38.9 (5.8) | 36.8 (6.4)

54. Secondary Outcome: Social Assuredness
Description: as for outcome 53
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.1 [-0.1 to 2.4] | 1.5 [0.3 to 2.7]

55. Secondary Outcome: Social Assuredness
Description: as for outcome 53
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.1 [-0.1 to 2.4] | 1.1 [-0.2 to 2.3]

56. Secondary Outcome: Social Assuredness
Description: as for outcome 53
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.9 [-0.4 to 2.2] | 1.8 [0.6 to 3.0]

57. Secondary Outcome: Physical Activity-International Physical Activity Questionnaire (IPAQ)
Description: Self-reported MVPA in bouts of 10 minutes or higher was measured using questions adapted from the International Physical Activity Questionnaire (IPAQ). The IPAQ is a nine-item instrument addressing days/week and minutes/day spent on physical activity in the past 7 days.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 61.8 (58.6) | 65.6 (87.5)

58. Secondary Outcome: Physical Activity-International Physical Activity Questionnaire (IPAQ)
Description: as for outcome 57
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 89.6 [54.3 to 124.8] | 42.7 [8.2 to 77.1]

59. Secondary Outcome: Physical Activity-International Physical Activity Questionnaire (IPAQ)
Description: as for outcome 57
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 91.0 [55.7 to 126.3] | 60.2 [25.9 to 94.6]

60. Secondary Outcome: Physical Activity-International Physical Activity Questionnaire (IPAQ)
Description: as for outcome 57
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: minutes per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
minutes per week | 30.5 [-5.4 to 66.5] | 28.4 [-6.2 to 63.0]

61. Secondary Outcome: Satisfaction With Intervention
Description: Participants will rate their overall satisfaction with the intervention on 7 point scale (7=completely satisfied, 1= completely dissatisfied).
Time Frame: 9 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 83 | 87
units on a scale | 2.2 [1.9 to 2.5] | 2.7 [2.4 to 3.0]

62. Secondary Outcome: Satisfaction With Intervention
Description: as for outcome 61
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 83 | 87
units on a scale | 2.3 [2.0 to 2.6] | 2.6 [2.3 to 2.9]

63. Secondary Outcome: Satisfaction With Intervention
Description: as for outcome 61
Time Frame: 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 83 | 87
units on a scale | 2.4 [2.1 to 2.7] | 2.5 [2.3 to 2.8]

64. Secondary Outcome: Frequency of Home Practice
Description: Participants will report the number of days per week they were able to practice skills taught in the program
Time Frame: 9 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: days per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 83 | 87
days per week | 4.3 [3.8 to 4.8] | 3.4 [2.9 to 3.9]

65. Secondary Outcome: Frequency of Home Practice
Description: Participants will report the number of days per week they were able to practice skills taught in the program
Time Frame: 26 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: days per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 83 | 87
days per week | 3.1 [2.6 to 3.5] | 3.0 [2.5 to 3.4]

66. Secondary Outcome: Frequency of Home Practice
Description: Participants will report the number of days per week they were able to practice skills taught in the program
Time Frame: 52 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: days per week
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 83 | 87
days per week | 3.2 [2.7 to 3.7] | 2.5 [2.1 to 3.0]

67. Secondary Outcome: Pain-11 Box Numerical Rating Scale
Description: An 11-box numerical rating scale (0=no pain, 10 = worst pain possible) for average back, neck, upper extremity, and lower extremity pain in the past week. The highest score for the assessed body regions was used for analysis.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 3.4 (2.3) | 3.3 (2.4)

68. Secondary Outcome: Pain-11 Box Numerical Rating Scale
Description: as for outcome 67
Time Frame: Change score: 9 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.4 [-0.1 to 0.9] | 1.0 [0.5 to 1.4]

69. Secondary Outcome: Pain-11 Box Numerical Rating Scale
Description: as for outcome 67
Time Frame: Change score: 26 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 0.9 [0.4 to 1.4] | 0.8 [0.3 to 1.2]

70. Secondary Outcome: Pain-11 Box Numerical Rating Scale
Description: as for outcome 67
Time Frame: Change score: 52 weeks - baseline
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
units on a scale | 1.0 [0.5 to 1.4] | 0.7 [0.2 to 1.2]

71. Secondary Outcome: Telehealth Usability Questionnaire
Description: Participant views of the remote intervention platform (Zoom video-conferencing system) were assessed using the Telehealth Usability Questionnaire (TUQ). The TUQ assesses usability with 21 questions rated on a 1 to 7 scale. The overall score is an average of all items with higher scores indicating higher usability of the telehealth system.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 45 | 43
units on a scale | 6.1 (0.7) | 5.9 (0.8)

72. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt uncomfortable with the facilitators. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A lower score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 46 | 43
units on a scale | 2.9 (2.6) | 1.9 (2.0)

73. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt uncomfortable with certain participants in the group. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A lower score indicates a higher bond with the group.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 46 | 43
units on a scale | 1.7 (1.4) | 2.0 (1.2)

74. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI task sub-scale asking participants how often they felt confused by what they were being asked to do in the sessions. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A lower score indicates a higher task alliance with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 46 | 43
units on a scale | 1.7 (1.1) | 2.0 (1.2)

75. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt the facilitators liked them. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A higher score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 45 | 43
units on a scale | 5.8 (1.6) | 6.0 (1.5)

76. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt the facilitators were genuinely concerned for their welfare. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A higher score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 45 | 43
units on a scale | 6.7 (0.8) | 6.6 (0.8)

77. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt the facilitators respected them. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A higher score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 46 | 43
units on a scale | 6.6 (0.9) | 6.8 (0.7)

78. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt the facilitators appreciated them. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A higher score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 45 | 43
units on a scale | 6.2 (1.3) | 6.2 (1.5)

79. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt confident the facilitators could help them if needed. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A higher score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 46 | 43
units on a scale | 6.4 (1.1) | 6.4 (1.2)

80. Secondary Outcome: Working Alliance Inventory (WAI)
Description: Question from the WAI bond sub-scale asking participants how often they felt their relationship with the facilitators was very important to them. Responses were recorded on a 1 to 7 scale with 1= Never and 7 = Always. A higher score indicates a higher bond with the facilitator.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 45 | 43
units on a scale | 5.0 (1.9) | 5.3 (1.8)

81. Secondary Outcome: Covid -19 Impact on Physical Activity
Description: Impact of COVID-19 on physical activity was assessed on a 5-item scale (1= substantially less physically active to 5 = substantially more physically active). The number of participants with reduced physical activity due to COVID-19 is reported.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 47 | 45
Participants | 42 | 42

82. Secondary Outcome: Covid -19 Impact on Physical Activity
Description: as for outcome 81
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 69 | 70
Participants | 54 | 52

83. Secondary Outcome: Covid -19 Impact on Physical Activity
Description: as for outcome 81
Time Frame: 26 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 68 | 70
Participants | 49 | 49

84. Secondary Outcome: Covid -19 Impact on Physical Activity
Description: as for outcome 81
Time Frame: 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 77 | 85
Participants | 64 | 67

85. Secondary Outcome: Number of Participants Completing Qualitative Assessment of Barriers to Intervention
Description: The number of participants completing qualitative, open ended assessments exploring dislikes and barriers to participation in the intervention.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
Participants | 83 | 84

86. Secondary Outcome: Number of Participants Completing Qualitative Assessment of Facilitators to Intervention
Description: The number of participants completing qualitative, open ended assessment exploring likes and facilitators to participation in the intervention.
Time Frame: 9 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
Number analyzed (Participants) | 86 | 90
Participants | 83 | 84

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the 1 year trial period.
Description: Adverse events (AEs) were monitored using active and passive surveillance. Participants were asked about the occurrence of potential AEs during all visits and surveys. In addition, participants were instructed to report adverse events to staff if they occurred. An independent safety monitor from the DSMB was responsible for classifying adverse events. Except for death, only adverse events classified as possibly, probably, or definitely related to the interventions are reported.
Arm/Group | Mindful Movement | Keys to Health & Wellbeing
All-Cause Mortality (participants affected / at risk) | 1/86 | 0/90
Serious Adverse Events (participants affected / at risk) | 7/86 | 6/90
Other Adverse Events (participants affected / at risk) | 40/86 | 51/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindful Movement (N=86) | Keys to Health & Wellbeing (N=90)
Cardiac conditions (e.g., atrial fibrillation, heart failure) (Cardiac disorders) | 1 (1) | 2 (2)
Hospitalization: Pseudosepsis (Vascular disorders) | 1 (1) | 0 (0) — Hospitalization for pseudosepsis following injection for increased knee pain with swelling
Hospitalization: Infection (COVID-19 or other) (Infections and infestations) | 0 (0) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 1 (1)
Hospitalization: Renal or Urinary disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hospitalization: Fracture or Dislocation (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hospitalization: Joint Replacement (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hospitalization: Vertigo or Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Amyloidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindful Movement (N=86) | Keys to Health & Wellbeing (N=90)
Increased pain (Musculoskeletal and connective tissue disorders) | 21 (23) | 24 (26) — Increase in musculoskeletal pain
Increased sadness, anxiousness, loneliness, or disturbing memories (Psychiatric disorders) | 18 (20) | 18 (18)
Increased fatigue (General disorders) | 3 (3) | 5 (5)
Infection (COVID-19 or other) (Infections and infestations) | 10 (10) | 16 (18)
Vertigo or Syncope (Nervous system disorders) | 2 (2) | 5 (6)

LIMITATIONS AND CAVEATS:
The interventions were transitioned to remote delivery as the trial was ongoing due to the COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT03929393/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/93/NCT03929393/ICF_000.pdf